CLINICAL TRIAL: NCT04200118
Title: Epigenetic and Genetic Effects in Cancer Patients: Analysis Pre and After Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IVI Barcelona (Other)
Responsible Party: Sponsor
Other Study IDs: 1901-BCN-011-MQ
Record Dates: First submitted 2019-12-04; First posted 2019-12-16 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-07

CONDITIONS: Male Infertility; Cancer; Epigenetic Disorder
Keywords: Sperm DNA fragmentation; Sperm epigenetics; Testicular cancer
MeSH Terms: conditions — Infertility, Male; Neoplasms; Testicular Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — non intervention

SUMMARY:
The prognosis in cancer patients has improved over the years. Survivor rates have increased significantly, and paternity has become an important concern in more than 50% of young male survivors. Sperm cryopreservation before cancer treatment is highly recommendable in these patients, as a strategy to preserve their fertility due to is not possible to predict how the chemo or radiotherapy treatment will affect the spermatogenesis.

The objective of this study is to evaluate if sperm after an antineoplastic treatment can be safely used. To determine the possible effects of oncological treatments in the spermatogenesis, three parameters will be analyzed, aneuploidy frequencies, DNA fragmentation in single and double-strand breaks and methylation levels to determine epigenetic changes before and after the therapy.

If cancer treatment affect sperm genetic integrity, it would have a clinical impact in the offspring of these patients. Identify the different side effects of antineoplastic treatments in DNA sperm will provide a clinical improvement in order to select the best sperm sample in an IVF treatment and it will facilitate genetic counseling

ELIGIBILITY:
Inclusion Criteria:

Patients with previous history of cancer Patients with several sperm samples cryopreserved to be able to thaw a part without damaging their future options, in case they need them.

Patients treated with chemotherapy and/or radiotherapy Patients have finished their oncological treatment. Patints recovered spermatogenesis after the oncological treatment to be able to obtain a sperm sample.

Exclusion Criteria:

Patients with only one sperm sample cryopreserved Patients that are not be able to obtain a fresh sample post treatment Patients with less than 3 million sperm per milliliter

Ages: 18 Years to 65 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Sperm samples before treatment will be used as a control
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-29 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Epigenetic profile of the patient | 3 months
  The epigenetic analysis will be performed in the laboratories of the company "Sequentia Biotech". The treatment of denatured DNA with sodium bisulfite will be carried out, causing the demining of the cytosine not methylated, preserving the integrity of the Metilcitosines. After DNA sequencing, treated with bisulfite, the methylation state can be inferred directly from the readings aligned against a reference genome: an unmodified cytosine will indicate the existence of methylation in that position, while A thymine (result of PCR amplification after demining) will mean the existence of a non-methylated cytosine. The methylation values will be calculated with the MethylDackel software and the statistical analysis with R package bsseq.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Ivi Barcelona, Barcelona
  - IVI Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided